CLINICAL TRIAL: NCT04141046
Title: LUPUS Brain: Transcranial Alternating Current Stimulation (tACS) to Target the Neurophysiology of Depression, Cognitive Deficits, and Pain in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: LUPUS Brain: tACS to Target the Neurophysiology of Depression, Cognitive Deficits, and Pain in Patients With SLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to end of funding period.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19-0763
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-05

CONDITIONS: Systemic Lupus Erythematosus; Depression
Keywords: Systemic lupus erythematosus; Lupus; SLE; Depression; Pain; Brain fog; Mood
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Depression; Pain; Mental Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research team and the participants will not know the intervention assignment until data is un-blinded for analysis.
  The Principal Investigators (PI) and Co-Investigators (Co-I) will be blinded since they may be outcome assessors and/or sub-specialty care providers for some of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Sham Stimulation (Sham Comparator): This is a sham/placebo arm that receives some stimulation, mimicking the skin sensations associated with tACS to enhance success of patient blinding.
  Interventions: Device: XCSITE100 Stimulator - Active Sham
- Theta-tACS (Active Comparator): This arm targets theta oscillations in the somatosensory cortex to see if there is a decrease in the experience of depression, pain, or brain fog in lupus patients.
  Interventions: Device: XCSITE100 Stimulator - Individualized theta-tACS
- Alpha-tACS (Experimental): This arm targets alpha oscillations in the somatosensory cortex to see if there is a decrease in the experience of depression, pain, or brain fog in lupus patients.
  Interventions: Device: XCSITE100 Stimulator - Individualized alpha-tACS

INTERVENTIONS:
Device: XCSITE100 Stimulator - Individualized theta-tACS — 20 second ramp-in and ramp-out with 40 minutes of stimulation for a total of 2440 seconds of stimulation
  Arms: Theta-tACS
Device: XCSITE100 Stimulator - Individualized alpha-tACS — 20 second ramp-in and ramp-out with 40 minutes of stimulation for a total of 2440 seconds of stimulation
  Arms: Alpha-tACS
Device: XCSITE100 Stimulator - Active Sham — 20 seconds of ramp-in to 40 seconds of 10 Hz tACS with a ramp out of 20 seconds for a total of 80 seconds of stimulation
  Arms: Sham Stimulation

SUMMARY:
The purpose of this study is to investigate the effects of a type of non-invasive transcranial alternating current stimulation (tACS) on patients diagnosed with systemic lupus erythematosus (SLE) who are experiencing depression.

Targeting depression in patients with SLE may provide benefit to these patients, as there is a clear relationship between chronic pain and depression. The investigators propose that a tACS stimulation montage that was previously used in depression could be beneficial to patients with SLE, resulting in reduced depression symptoms, thus resulting in reduced chronic pain and cognitive difficulties.

DETAILED DESCRIPTION:
At the initial session, consent will be obtained and eligibility will be determined.

Eligible participants will undergo a structural MRI as part of the screening process, then be randomized and have 5 consecutive daily, 40 minute stimulation sessions.

Participants will be randomly assigned to one of three groups: sham stimulation, individualized alpha-tACS (usually 8-12 Hz), or individualized theta-tACS (individualized alpha frequency minus 4 Hz). Participation will include 1 to 11 visits.

Neurophysiological measures will be taken before and after the stimulation sessions on the first and fifth days of the intervention, as well as the 2-week follow-up and 4-week follow-up visits. Psychiatric clinical assessments will be performed at baseline (Day 1 of stimulation), Day 5 of stimulation, and at both follow-up visits using the Hamilton Depression Rating Scale (HDRS17), the Hamilton Anxiety Rating Scale (HAM-A), the Inventory of Depression and Anxiety Symptoms (IDAS), and the Comparative Pain Scale Chart. All participants will also be asked to complete self-report surveys via REDCap at a 3-month time point measured from completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years
* Meets SLE diagnosis criteria
* Low suicide risk
* Not experiencing a manic episode
* Stable on all SLE and psychiatric medications for 6 weeks prior to screening
* Capacity to understand all relevant risks and potential benefits of the study

Exclusion Criteria:

* Drug-induced SLE and any other rheumatologic or autoimmune disease diagnosis (except for Sjogren's syndrome and mixed connective tissue disease)
* Medical illness (unstable cardiac disease, AIDS, liver or renal impairment, or malignant disease within 5 years before screening visit) or treatment of same that could interfere with study participation
* Neurological disorders, including but not limited to history of seizures (except childhood febrile seizures and electroconvulsive therapy induced seizures), dementia, history of stroke, Parkinson's disease, multiple sclerosis, cerebral aneurysm; History of moderate to severe traumatic brain injury (TBI); Frequent or severe migraines in the past 30 days before the screening visit
* History of positive hepatitis B, hepatitis C antibody, HIV antibody/antigen; Opportunistic infection in the 12 weeks before initial study dosing OR currently undergoing treatment for a chronic opportunistic infection (TB, pneumocystis pneumonia, cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacteria); Acute OR chronic infection requiring hospitalization in the 30 days before screening visit AND/OR administration of parenteral (IV or IM) antibacterial, antiviral, antifungal, or anti-parasitic agents in the 30 days before screening visit
* Have received intravenous glucocorticoids at a dosage of ≥ 500mg daily within the past month; Current use of benzodiazepines or anti-epileptic drugs
* History of thrombophlebitis or thromboembolic disorders (e.g., blood clots) or serious adverse reactions to blood draws
* Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnosis of alcohol of substance abuse (other than nicotine) within the last month or a DSM-IV diagnosis of alcohol or substance dependence (other than nicotine) within the last 6 months; Prior or current diagnosis of bipolar disorder, manic episodes, hypomanic episodes, or mixed episodes; Prior or current diagnosis of a psychotic disorder
* Prior brain surgery; Any brain devices/implants, including cochlear implants and aneurysm clips or other factors that are contraindicated for undergoing an MRI
* Pregnancy, nursing, or if female and fertile, unwilling to use appropriate birth control measures during study participation
* Concurrent medical condition or treatment for a medical disorder that, in the opinion of the investigator, could confound interpretation of results or affect the patient's ability to fully participate in the study.
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study
* Non-English speakers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saira Z Sheikh, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data sharing requests will become available starting from 9 to 36 months following publication.
Access Criteria: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the interested investigator provides a (1) written request to the PI, (2) approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and (3) executes a data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were randomized to the Theta-tACS arm.
Groups:
- Sham Stimulation: This is a sham/placebo arm that receives some stimulation, mimicking the skin sensations associated with Transcranial Alternating Current Stimulation (tACS) to enhance success of patient blinding.
  XCSITE100 Stimulator - Active Sham: 20 seconds of ramp-in to 40 seconds of 10 Hz tACS with a ramp out of 20 seconds for a total of 80 seconds of stimulation
Period: Overall Study
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Started | 1 | 0 | 3
Completed | 1 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were randomized to the Theta-tACS arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS | Total
Number analyzed (Participants) | 1 | 0 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0 | 0
  Between 18 and 65 years | 1 |  | 3 | 4
  >=65 years | 0 |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 3 | 4
  Male | 0 |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0 | 0
  Not Hispanic or Latino | 1 |  | 3 | 4
  Unknown or Not Reported | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 0 | 0
  White | 1 |  | 3 | 4
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 |  | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Alpha Oscillation Power as Measured by RSEEG Recordings.
Description: Change in alpha oscillation power (8-12 Hz) will be measured between resting state electroencephalogram (RSEEG) recordings.
Time Frame: Day 1, Day 5
Population: No participants were randomized to the Theta-tACS arm.
Measure: Mean (Standard Deviation); unit: microvolts^2/Hz
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Number analyzed (Participants) | 1 | 0 | 3
microvolts^2/Hz | 0.146 |  | -0.015 (0.11)

2. Secondary Outcome: Change in Correlation Between the IDAS Score and Alpha Oscillation Power (as Measured by Resting State EEG Recordings).
Description: The Inventory of Depression and Anxiety Symptoms (IDAS) Scale is a 10 symptom scale (General depression, Suicidality, Lassitude, Insomnia, Appetite Loss, Appetite Gain, Ill Temper, Well-Being, Panic, Social Anxiety, and Traumatic Intrusions) used to assess depression and anxiety related disorders. The scale ranges from 1 to 5 with 1 equal to "not at all" and 5 equal to"extremely". Higher scores indicate a greater experience of a given symptom.
Time Frame: Day 1, Day 5
Population: Insufficient data were collected to validly calculate a correlation as stated in the statistical analysis plan.
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in Correlation Between the PANAS Score and Alpha Oscillation Power (as Measured by Resting State EEG Recordings).
Description: The Positive and Negative Affect Schedule (PANAS) will be used to measure positive and negative emotion. This 20-item self-reported survey will measure 10 positive and 10 negative affective states. Positive affect score ranges from 10-50 and higher scores indicate a greater positive affect. Negative affect scores range from 10-50 with higher scores indicating a greater negative affect.
Time Frame: Day 1, Day 5
Population: Insufficient data were collected to validly calculate a correlation as stated in the statistical analysis plan.
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in Correlation Between the Comparative Pain Scale Score and Alpha Oscillation Power (as Measured by Resting State EEG Recordings).
Description: The Comparative Pain Scale score will assess for self-reported pain. The scale ranges from 0 to 10, with 0 equal to "pain free" and 10 equal to "unmanageable, unspeakable". Higher scores reflect a higher severity of self-reported pain.
Time Frame: Day 1, Day 5
Population: Insufficient data were collected to validly calculate a correlation as stated in the statistical analysis plan.
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change in Correlation Between the Short Form Health Survey (SF-36) Score and Alpha Oscillation Power (as Measured by Resting State EEG Recordings).
Description: The 36-Item Short Form Health Survey (SF-36) measures general health using 36 questions. There are 8 individual health "domains" or categories that each receive their own score, and from these 8 individual scores an overall score can be obtained. Overall scores can range from 0-100, with higher scores indicating better overall health.
Time Frame: Screening, 4 week
Population: Insufficient data were collected to validly calculate a correlation as stated in the statistical analysis plan.
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in Correlation Between the FSMC Score and Alpha Oscillation Power (as Measured by Resting State EEG Recordings).
Description: The Fatigue Scale for Motor and Cognitive Functions (FSMC) will measure self-reported levels of physical and mental fatigue. This 20-item survey will measure 10 motor fatigue items and 10 cognitive fatigue items. The scale ranges from 1 to 5 with 1 equal to "does not apply at all" and 5 equal to "applies completely". Total scores can range from 20 to 100 with higher scores indicating worse fatigue.
Time Frame: Day 1, Day 5
Population: Insufficient data were collected to validly calculate a correlation as stated in the statistical analysis plan.
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change in Correlation Between the PCS Score and Alpha Oscillation Power (as Measured by Resting State EEG Recordings).
Description: The Pain Catastrophizing Scale (PCS) will assess for self-reported pain. The survey consists of 13 items with a 5-point scale, where 0 equals"not at all" and 4 equals "all the time". Total scores can range from 0 to 52 with higher scores indicating a greater frequency in which individuals experience pain-related thoughts and feelings.
Time Frame: Day 1, Day 5
Population: Insufficient data were collected to validly calculate a correlation as stated in the statistical analysis plan.
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change in Correlation Between the YMRS Score and Alpha Oscillation Power (as Measured by Resting State EEG Recordings).
Description: The Young Mania Rating Scale (YMRS) will assess for manic symptoms at baseline and over the period of the study. The 11 item scale ranges from 0 to 56 with higher scores indicating more severe manic symptoms.
Time Frame: Day 1, Day 5
Population: Insufficient data were collected to validly calculate a correlation as stated in the statistical analysis plan.
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change in Correlation Between the HDRS17 Score and Alpha Oscillation Power (as Measured by Resting State EEG Recordings).
Description: The Hamilton Depression Rating Scale (HDRS17) will assess for the severity of depressive symptoms in the patients. The scale ranges from 0 to 52 with higher scores indicating a greater severity of depressive symptoms.
Time Frame: Day 1, Day 5
Population: Insufficient data were collected to validly calculate a correlation as stated in the statistical analysis plan.
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Change in Correlation Between the HAM-A Score and Alpha Oscillation Power (as Measured by Resting State EEG Recordings).
Description: The Hamilton Anxiety (HAM-A) scale will assess for the severity of anxiety symptoms. The scale ranges from 0 to 30 with higher scores indicating greater anxiety.
Time Frame: Day 1, Day 5
Population: Insufficient data were collected to validly calculate a correlation as stated in the statistical analysis plan.
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
Number analyzed (Participants) | 0 | 0 | 0

11. Other Pre Specified Outcome: Change in Correlation Between Frontal Midline Alpha and Theta Activity (as Measured From EEG Recordings) and Accuracy at Cognitive Tasks Tasks.
Description: Participants will complete various tasks paired with electroencephalogram (EEG) recordings to assess physiological changes. Participants will be asked to perform sustained attention, selective attention, and working memory tasks with EEG recordings.
Time Frame: Day 1, Day 5
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in the WHODAS 2.0 Score.
Description: The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) will assess for co morbid disabilities. This 12-item survey ranges from 0 to 4 with 0 being "none" and 4 being "extreme or cannot do". Total scores can range from 0 to 48 with higher scores lower levels of social functioning.
Time Frame: Day 1, 3 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through study completion, a total of approximately 3 months.
Description: No participants were randomized to the Theta-tACS arm. In addition to the standard ClinicalTrials.gov Serious Adverse Event definition, the study also defined an adverse event of grade 3 or higher as determined by the U.S. Department of Health and Human Services' Common Terminology Criteria for Adverse Events (CTCAE Version 5.0 Published: November 27th, 2017) as a Serious Adverse Event.
Arm/Group | Sham Stimulation | Theta-tACS | Alpha-tACS
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 2/3
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Stimulation (N=1) | Theta-tACS (N=0) | Alpha-tACS (N=3)
Vasovagal response (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Newly Diagnosed Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Lesion present at screening visit
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Stimulation (N=1) | Theta-tACS (N=0) | Alpha-tACS (N=3)
Laceration from pet claw (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Elevated Blood pressure (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated Urine Protein (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT04141046/Prot_SAP_000.pdf